CLINICAL TRIAL: NCT02636166
Title: Project-0027 Lay User Usage Study
Brief Title: Project-0027. Lay User Usage Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SPD Development Company Limited (Industry)
Collaborators: Illingworth Research Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PROTOCOL-0772
Record Dates: First submitted 2015-10-20; First posted 2015-12-21 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-10

CONDITIONS: Pregnancy
Keywords: Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pregnancy test (Other): Clearblue investigational Pregnancy test
  Clearblue Marketed pregnancy test
  Professional pregnancy test
  Interventions: Other: Clearblue Investigational Pregnancy test; Other: Professional pregnancy test; Other: Clearblue Marketed Pregnancy test

INTERVENTIONS:
Other: Clearblue Investigational Pregnancy test — Clearblue Investigational Pregnancy test
Other: Professional pregnancy test — Alere Professional use pregnancy test
Other: Clearblue Marketed Pregnancy test — Clearblue Marketed Pregnancy test

SUMMARY:
Study volunteers will be required to conduct a home pregnancy test (HPT) at the trial centre and provide a sample of urine from the same void for further testing.

Volunteers will then complete a product usage questionnaire and leaflet comprehension questionnaire at site.

Follow-up information will be required from all volunteers as both additional urine sample(s) and pregnancy information to establish true pregnancy status at the study visit.

DETAILED DESCRIPTION:
Eligible volunteers will be recruited into the study and provide informed consent. Volunteers will then test their urine sample with the investigational HPT according to the device Instructions for use and record their result onto the results sheet. A sample of urine from the same void will be obtained for further testing by the study technicians.

The technician will then test the volunteer's sample with a second investigational HPT, a professional use pregnancy test and a Clearblue Digital HPT, the results of which will be used to provide the volunteer with her pregnancy test result. During technician testing, the volunteer will complete the device usability and leaflet comprehension questionnaires.

At the end of the study visit, all volunteers will be provided with materials to allow follow-up for the determination of pregnancy status.

The majority of volunteers will be requested to provide one additional urine sample, collected 2 days after the study visit. If early pregnancy is suspected the volunteer will be requested to provide an additional 7 daily urine samples following the study visit. All volunteers will be required to provide details of pregnancy status (documented menses or pregnancy confirmation by health care professional) after the study visit.

True pregnancy status will be determined by laboratory tests and clinical information. The study will continue until a minimum of 300 pregnant and 300 not pregnant volunteers have completed the study.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged 18 or over
* Willing to conduct a personal pregnancy test and reveal their pregnancy status
* Willing to give informed consent

Exclusion Criteria:

* Currently or previously employed by SPD Development Company Ltd. (SPD), Alere, Unipath, Procter and Gamble (P&G), or affiliates.
* Has an immediate relative* currently or previously employed by SPD, Alere, Unipath or P&G or affiliates
* Previously used the investigational HPT within the last six months
* Healthcare professionals (HCP's) with professional experience either using lateral flow based devices or conducting near patient testing
* Confirmed to be pregnant by a healthcare professional and beyond the first trimester
* Taken a hormonal preparation containing human chorionic gonadotropin (hCG) in the last month, e.g. Pregnyl®

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 943 (Actual)
Dates: Start 2015-07; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of participants recording the correct pregnancy test result when testing their own urine sample with the investigational HPT referenced to confirmed pregnancy status | 3 months
  The accuracy of the investigational HPT in volunteer hands compared to pregnancy status

SECONDARY OUTCOMES:
Number of participants recording the same pregnancy test result as a laboratory technician when testing their own urine sample with the investigational HPT. | 3 months
  The agreement between volunteer and technician results using the investigational HPT
Number of participants recording a false positive or false negative pregnancy test result when testing their own urine sample with the investigational HPT referenced to confirmed pregnancy status. | 3 months
  The estimated sensitivity and specificity of the investigational HPT
Calculation of the level of certainty a user can have if the device gives a pregnant (positive predictive value (PPV)) or not pregnant result (Negative predictive value(NPV)). | 3 months
  The estimated NPV and PPV of the investigational HPT
Number of participants correctly answering questions about the product when referencing the instructions for use (IFU) leaflet. | 3 months
  Volunteer leaflet comprehension of the IFU
Participants opinion on using the product. | 3 months
  Volunteer usability of the IFU

CONTACTS AND LOCATIONS:
Overall Officials: Juliet Hulse, Principal Investigator — Illingworth Research Ltd
Locations (1):
- Illingworth Research Ltd, Macclesfield, Chester, United Kingdom